CLINICAL TRIAL: NCT03749538
Title: Acute Transcranial Direct Current Stimulation in Patients With Systemic Autoimmune Myopathies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Professor, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MYO-HCFMUSP-06
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Myopathy; Neurologic Manifestations; ElectroPhys: Myopathy
MeSH Terms: conditions — Muscular Diseases; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled study with application or not of a transcranial current stimulation session in patients with systemic autoimmune myopathies.
Who Masked: Participant, Investigator
Masking Description: Double-blind study to transcranial current stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial direct current stimulation (Experimental): Transcranial direct current stimulation session: the energy of the anode (transcranial current stimulation) will have as its source a battery-powered DC generator and will be exerted by two electrodes measuring 5x7cm and attached to the head. The electrodes will be located of the primary motor cortex. The electrode with positive charge (anode) will be positioned at contralateral to the dominant limb and the negative charged electrode will be positioned in the supraorbital region ipsilateral to the dominant limb. The active current of direct transcranial stimulation will be applied with the intensity of electric current of 2mA and density of 0.057 mA/cm2 with duration of 20 minutes. During the session, patients will remain seated. Number of sessions: three times, once per day.
  Interventions: Other: Transcranial direct current stimulation session.
- Placebo (Placebo Comparator): This group will not receive a transcranial direct current stimulation session.
  Interventions: Other: Transcranial direct current stimulation session.

INTERVENTIONS:
Other: Transcranial direct current stimulation session. — Patients with systemic autoimmune myopathies will receive or not acute transcranial direct current stimulation session.

SUMMARY:
Systemic autoimmune myopathies are a heterogeneous group of rheumatic diseases that primarily affect the skeletal muscles. The transcranial direct current stimulation technique has been frequent, for example, in patients with ischemic stroke or for the optimization of muscular performance in athletes. However, to date, there are no studies evaluating this technique in patients with systemic autoimmune myopathies. Therefore, the main objective of the present prospective, randomized, double-blind, placebo-controlled study is to evaluate the safety and efficacy of the application of acute transcranial current stimulation session in patients with systemic autoimmune myopathies.

DETAILED DESCRIPTION:
Currently, there are no studies evaluating the transcranial current stimulation technique in patients with systemic autoimmune myopathies. Therefore, the main objective of the present prospective, randomized, double-blind, placebo-controlled study is to evaluate the safety and efficacy of the application of acute transcranial direct current stimulation session in patients with systemic autoimmune myopathies.

ELIGIBILITY:
Inclusion Criteria:

* Classification criteria - EULAR/ACR 2017
* Classification critera - Connors et al.
* Objective muscle limb weakness

Exclusion Criteria:

* Neoplasia
* Using heart pacemarker
* Using visceral metalic clips
* Infections (HIV, HTLV-1, Hepatitis, etc)
* Pregnance
* Previous historical of convulsions or epilepsies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events [safety and tolerability] | After 30 minutes of transcranial stimulation.
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)
Frequency of treatment-emergent adverse events [safety and tolerability] | After 8 weeks of transcranial stimulation.
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration)

SECONDARY OUTCOMES:
Myositis Disease Activity Assessment Visual Analogue Scales (MYOACT) | 3 times: (a) within 30 minutes before stimulation. Then, after (b) 3 weeks and (c) 8 weeks after stimulation.
  This partially validated tool measures the degree of disease activity of extra-muscular organ systems and muscle. The questionnaire is a series of physician's assessments of disease activity. Score ranges: 0 (best) - 60 (worst).
Serum levels of Muscle enzymes | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation.
  This partially validated tool measures the serum activities of at least 2 of the 4 muscle-associated enzymes including creatine phosphokinase (CK), the transaminases (ALT, AST), lactate dehydrogenase (LD) and aldolase. The reference range value of each muscle enzyme will depend on the laboratory anaysis (kits). International Unit: U/L.
Health Assessment Questionnaire (HAQ) | 3 times: (a) within 30 minutes before stimulation. Then, after (b) 3 weeks and (c) 8 weeks after stimulation
  Especific questionnaire (health assessment questionnaire). Pontuaction 0.00 (best) - 3.00 (worst)
Manual Muscle Testing (MMT) | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation.
  This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies. Pontuaction: 0 (worst) - 80 (best)
Patient Global Activity | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation.
  This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale. Pontuaction: 0 (best) - 10 (worst)
Physician Global Activity | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation.
  This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. visual analogue scale. Pontuaction: 0 (best) - 10 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, Principal Investigator — Universidade de Sao Paulo - Rheumatology Division
Locations (1):
- Samuel K Shinjo, São Paulo, Brazil